CLINICAL TRIAL: NCT01828021
Title: A Single Arm, Open-Label, Phase 2 Study of MGAH22 (Fc-optimized Chimeric Anti-HER2 Monoclonal Antibody) in Patients With Relapsed or Refractory Advanced Breast Cancer Whose Tumors Express HER2 at the 2+ Level by Immunohistochemistry and Lack Evidence of HER2 Gene Amplification by FISH
Brief Title: Phase 2 Study of the Monoclonal Antibody MGAH22 (Margetuximab) in Patients With Relapsed or Refractory Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGAH22-02
Record Dates: First submitted 2013-03-26; First posted 2013-04-10 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: HER2 2+; FISH non-amplified; Relapsed; Refractory; Advanced; Margetuximab; MGAH22
MeSH Terms: conditions — Breast Neoplasms; Recurrence | interventions — margetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- margetuximab (Experimental): Monotherapy of Anti-HER2 monoclonal antibody
  Interventions: Biological: Margetuximab

INTERVENTIONS:
Biological: Margetuximab — Anti-HER2 monoclonal antibody
  Other Names: MGAH22

SUMMARY:
The purpose of this study is to determine if margetuximab is effective in the treatment of certain patients with relapsed or refractory advanced breast cancer.

DETAILED DESCRIPTION:
In the pivotal study that established that Herceptin® was highly effective when added to standard chemotherapy in the front-line treatment of women with HER2 positive metastatic breast cancer, benefit appeared to accrue to those patients whose tumors expressed the HER2 oncoprotein at the 3+ level by immunohistochemistry (IHC) or those patients whose tumors demonstrated evidence of HER2 gene amplification by fluorescence in situ hybridization (FISH) testing. Similarly, when Herceptin® was used as a single therapy in women with metastatic breast cancer that had progressed following cytotoxic chemotherapy, 3+ overexpression of HER2, but not 2+ expression, was associated with response to treatment. These and other studies have led to the recommendation that Herceptin® should be administered to patients with breast cancer whose tumors exhibit 3+ overexpression or gene amplification. This study will evaluate whether treatment of patients with tumors that would not be expected to respond to Herceptin® therapy, namely those that lack HER2 gene amplification and express the oncoprotein at the 2+ level by IHC, may benefit from the use of the anti-HER2 monoclonal antibody, MGAH22. If 5 or more responses are seen in 41 evaluable patients, then further clinical development of margetuximab will be justified.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive carcinoma of the breast
* Treatment with at least two prior systemic therapies for advanced (unresectable locoregional or metastatic) disease
* Evidence of HER2 oncoprotein expression at the 2+ level by central laboratory. Patients whose tumors exhibit 2+ staining by IHC are eligible for the study.
* Patients whose tumors score 1+ by conventional IHC, are non-amplified by FISH testing, and whose tumors score > or = 10.5 by HERmark® testing, are eligible for the study.
* Evidence of lack of HER2 oncogene amplification as determined by FISH testing by central laboratory
* Performance Status of 0 or 1
* Life expectancy at least 6 months
* Measurable disease (by RECIST 1.1)
* Acceptable laboratory parameters and organ reserve
* Baseline left ventricular ejection fraction > or = 50%
* Anti-cancer therapy (including conventional cytotoxic chemotherapy and/or biological therapy) and radiotherapy must be completed and any associated toxicities resolved to </= Grade 1 levels or baseline levels and at least 2 weeks must have elapsed before enrollment. Treatment with monoclonal antibodies must be completed at least 14 days before entry. Must have completed immunosuppressive medications or vaccinations before enrollment.
* Patients who are estrogen receptor+ and/or progesterone receptor+ and who are receiving anti-hormone therapy for at least three months may continue to receive such therapy during the course of the trial
* Eighteen (18) years of age or older

Exclusion Criteria:

* Major surgery or trauma within 4 weeks
* Known hypersensitivity to murine or recombinant proteins, polysorbate 80, or any excipient contained in the margetuximab drug formulation
* Second primary malignancy that has not been in remission for more than 3 years
* History of active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 14 days
* History within 3 months of deep vein thrombosis, pulmonary embolism, or stroke
* Symptomatic or untreated central nervous system (CNS) metastatic disease. Patients with previously treated CNS metastatic disease which has been stable for at least 56 days are eligible
* Requirement, at time of study entry, for concurrent steroids > 10 mg/day of oral prednisone or the equivalent, except steroid inhaler, nasal spray, or ophthalmic solution
* Serious medical condition that would impair the ability to receive or tolerate margetuximab; dementia or altered mental status that would preclude provision of informed consent
* Uncontrolled hypertension, heart disease including history of congestive heart failure, history of myocardial infarction, angina pectoris requiring medication, clinically significant valvular heart disease, high risk arrhythmias, or disease corresponding to New York Heart Association class III or IV.
* Significant pulmonary compromise
* Have previously been exposed to MGAH22 in this or any other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Florida Cancer Research Institute, Plantation, Florida
  - Indiana University, Indianapolis, Indiana
  - Tufts Cancer Center, Boston, Massachusetts
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nordstrom JL, Gorlatov S, Zhang W, Yang Y, Huang L, Burke S, Li H, Ciccarone V, Zhang T, Stavenhagen J, Koenig S, Stewart SJ, Moore PA, Johnson S, Bonvini E. Anti-tumor activity and toxicokinetics analysis of MGAH22, an anti-HER2 monoclonal antibody with enhanced Fcgamma receptor binding properties. Breast Cancer Res. 2011;13(6):R123. doi: 10.1186/bcr3069. Epub 2011 Nov 30. PMID 22129105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred at 6 US oncology centers -- 4 academic institutions and 2 clinical research centers, between May 2013 and November 2016.
Groups:
- Margetuximab: Monotherapy of Anti-HER2 monoclonal antibody
  Margetuximab: Anti-HER2 monoclonal antibody
  Margetuximab was administered by IV infusion at a dose of 6.0 mg/kg on Days 1, 8, and 15 of each 28-day cycle or or 15 mg/kg every 3 weeks of each 21-day cycle
Period: Overall Study
Arm/Group | Margetuximab
Started | 25
Completed | 0
Not Completed | 25
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 17
Not completed — Withdrawal by Subject | 2
Not completed — Ileal obstruction, unrelated | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of margetuximab
Arm/Group | Margetuximab
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status assesses how the disease affects the daily living abilities of the patient and how the disease is progressing or improving. The scale ranges from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead); therefore, lower numbers indicate better status.
  Participants
    Performance Status 0 | 14
    Performance Status 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Response based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria based on Cycle 2, Day 21 computed tomography (CT) scans. Response is categorized as complete response (CR): disappearance of all target lesions, confirmed at ≥ 4 weeks; partial response (PR): ≥ 30% decrease in target lesions from baseline, confirmed at ≥ 4 weeks; progressive disease (PD): ≥ 20% increase over smallest sum observed with an absolute increase of at least 5 mm, or appearance of new lesions; and stable disease (SD): neither PR or PD criteria met.
  A Simon two-stage design was planned in which an initial cohort of 21 patients was treated. If 2 or more responses (PR or CR) are seen at the first tumor re-evaluation on day 21 of Cycle 2, the study would be expanded to include up to 41 patients (20 additional patients in Cohort 2, the second stage of the study) in order to determine whether further development of the drug is warranted (5 or more responses in 41 evaluable patients).
Time Frame: Cycle 2, Day 21
Population: All patients with baseline tumor evaluation, received any amount of study drug, and had a tumor evaluation at Cycle 2 Day 21
Measure: Number; unit: participants
Arm/Group | Margetuximab
Number analyzed (Participants) | 22
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 6
  Progressive Disease | 12
  Not Done | 4

2. Secondary Outcome: Response Rate
Description: Response rate is the proportion of patients achieving a best response of complete response or partial response when such responses are confirmed at least 28 days after initial observation of response.
  Response based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria based on Cycle 2, Day 21 computed tomography (CT) scans. Response is categorized as complete response (CR): disappearance of all target lesions, confirmed at ≥ 4 weeks; partial response (PR): ≥ 30% decrease in target lesions from baseline, confirmed at ≥ 4 weeks; progressive disease (PD): ≥ 20% increase over smallest sum observed with an absolute increase of at least 5 mm, or appearance of new lesions; and stable disease (SD): neither PR or PD criteria met.
Time Frame: Day 49
Population: All patients with baseline tumor measurement, at least one dose of study drug, and Cycle 2 Day 21 tumor assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab
Number analyzed (Participants) | 22
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent until End of Study visit; average time on treatment was 35.6 days
Arm/Group | Margetuximab
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Margetuximab (N=25)
Ascites (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Margetuximab (N=25)
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 6
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Headache (Nervous system disorders) | 4
Neuropathy periphera (Nervous system disorders) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 5
Procedural nausea (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Ejection fraction decreased (Investigations) | 2
Lymphoctye count decreased (Investigations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No